CLINICAL TRIAL: NCT00181935
Title: Open-Label Comparative Study of Risperidone Versus Olanzapine for Mania in Preschool Children 4 to 6 Years of Age With Bipolar Spectrum Disorder
Brief Title: Risperidone Versus Olanzapine for Mania in Preschool Children 4 to 6 Years of Age With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2001-P-000422
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Bipolar Disorder; Mania
Keywords: bipolar disorder; preschoolers; risperdal; zyprexa
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: risperidone (Risperdal)
Drug: olanzapine (Zyprexa)

SUMMARY:
The objectives of this study are to study the safety, effectiveness, tolerability and dosing regimen of risperidone, and olanzapine, in the treatment of mania in Bipolar Disorder I and Bipolar II Disorder in preschool children over an 8 week period. We hypothesize that these atypical neuroleptics may be effective in treating pediatric mania, with a lower risk of extrapyramidal side effects.

DETAILED DESCRIPTION:
Risperidone and olanzapine are atypical neuroleptics marketed for the treatment of psychotic disorders in adults. These medicines are called atypical neuroleptics because of their unique pharmacological profile, which include both D2 and 5HT2 antagonistic effects. The combined dopaminergic and serotonergic activity seems to be associated not only with antipsychotic effects, but also with mood stabilizing, mood elevating and tardive dyskinesia. The anti-climactic effects of this class of drugs led to the recent FDA approval of olanzapine as monotherapy for adult bipolar disorder.

The study will consist of 8 week, open-label treatment period with random assignment to two determined treatment arms, risperidone or olanzapine. We plan to enroll 5 subjects for each arm. During the 8 weeks of treatment, patients will be seen at weekly intervals and receive study medication. At each week, measures of safety and efficacy will be obtained. Two teams of clinicians will see the patient at each visit. Team 1 will be the treating team, adjusting medication dosages and determining the safety of continuation in the study for the patient. Team 2 will be blind to the randomization status of the patient and will assess clinical improvement using the efficacy measures. For patients who have completed the 8-week acute phase without adverse event and have not responded to the medication they were assigned to will be allowed to then take part in additional 8-week trial with the other medication. At the end of the 8 weeks, patients who responded to their assigned treatment will be eligible to be enrolled and invited to participate in a separate10 month continuation study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 4-6 years of age.
2. Parent or legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
3. Patients and their legal representative must be considered reliable.
4. Each patient and his/her authorized legal representative must understand the nature of the study. The patient's authorized legal representative must sign an informed consent document.
5. Patient must have a diagnosis of bipolar I or bipolar II disorder and currently displaying an acute manic, hypomanic, or mixed episode (with or without psychotic features) according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kidd Schedule of Affective Disorders).
6. Patients must have an initial score on the Y-MRS total score of at least 15.
7. Patient must be able to participate in mandatory blood draws.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious, unstable illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease
3. Uncorrected hypothyroidism or hyperthyroidism.
4. History of severe allergies or multiple adverse drug reactions.
5. Non-febrile seizures without a clear and resolved etiology.
6. Leukopenia or history of leukopenia without a clear and resolved etiology.
7. Judged clinically to be at serious suicidal risk.
8. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol
9. History of intolerance or non-responder to risperidone, or olanzapine as determined by the principal investigator.
10. Treatment with nonreversible monoamine oxidase inhibitor within 2 weeks prior to Visit 2.
11. Current diagnosis of schizophrenia.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 2001-03; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
reduction in symptoms measured by
Young Mania Rating Scale
Mania Symptom Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States